CLINICAL TRIAL: NCT03041376
Title: Effect of Pedometer-Based Walking Intervention on Functional Capacity and Neurohumoral Modulation in Patients With Chronic Heart Failure With Preserved Ejection Fraction: a Multicenter Randomized Controlled Trial
Brief Title: Pedometer-Based Walking Intervention in Patients With Chronic Heart Failure With Preserved Ejection Fraction
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charles University, Czech Republic (Other)
Collaborators: General University Hospital, Prague (Other); Brno University Hospital (Other); University Hospital Olomouc (Other); University Hospital Hradec Kralove (Other); Tomas Bata Hospital, Czech Republic (Other)
Responsible Party: Principal Investigator, Jan Belohlavek, Ass. Prof., Charles University, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Walking in HFpEF
Record Dates: First submitted 2017-02-01; First posted 2017-02-02 (Estimated); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Diastolic Heart Failure
MeSH Terms: conditions — Heart Failure, Diastolic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Walking intervention (Experimental)
  Interventions: Behavioral: Walking intervention
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Walking intervention — The intervention will be delivered over a six-month period and will consist of: (1) an individualized pedometer-based walking program with weekly step goals, (2) regular visits to the clinic including face-to-face session with the physician, and (3) regular telephone calls with the research nurse in between the face-to-face contacts.
  Arms: Walking intervention

SUMMARY:
A multicenter randomized controlled trial, with follow-up at 6 and 12 months. Physically inactive participants with chronic heart failure with preserved or mid-range ejection fraction will be randomly assigned to intervention or control arms.

The six-month intervention will consist of an individualized pedometer-based walking program with weekly step goals, monthly face-to-face sessions with the physician, and monthly telephone calls with the research nurse. The intervention will be based on effective behavioral principles (goal setting, self-monitoring, personalized feedback).

The primary outcome is the change in 6-minute walk distance at 6 months. Secondary outcomes include changes in serum biomarkers levels, pulmonary congestion assessed by ultrasound, average daily step count measured by accelerometry, anthropometric measures, symptoms of depression, health-related quality of life, self-efficacy, and MAGGIC Risk Score.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of heart failure with preserved (HFpEF) or mid-range (HFmrEF) ejection fraction with New York Heart Association (NYHA) class II or III symptoms. The diagnosis requires the following conditions to be fulfilled:

   1. the presence of symptoms and/or signs of heart failure,
   2. left ventricular ejection fraction ≥50% (HFpEF) or 40-49% (HFmrEF),
   3. elevated levels of natriuretic peptides (BNP >35 pg/ml and/or NT-proBNP >125 pg/mL),
   4. objective evidence of other cardiac functional and structural alterations underlying heart failure.
2. Physically inactive, as determined by a question "As a rule, do you do at least half an hour of moderate or vigorous exercise (such as walking or a sport) on five or more days of the week?".

Exclusion Criteria:

1. Signs and symptoms of decompensated heart failure, uncontrolled arrhythmia or effort angina, severe or symptomatic aortic stenosis, persistent hypotension, recent shocks delivered by the automated implantable cardioverter defibrillator.
2. Co-morbid conditions that would affect adherence to trial procedures (e.g. inflammatory arthritis, active malignancy, renal disease requiring dialysis, uncontrolled diabetes, major depression or other significant psychiatric disorders, cognitive impairment, significant hearing or visual impairment).
3. Major surgery planned within the next 12 months.
4. Life expectancy shorter than 12 months.
5. Inability to walk from any reason.
6. Baseline six-minute walking distance >450 meters. Patients covering more than 450 meters in the baseline six-minute walk test (6MWT) are excluded due to a possible ceiling effect.
7. Pregnancy.
8. Failure to perform the 6MWT.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-04-11 (Actual); Primary Completion 2019-06-30 (Estimated); Study Completion 2020-01-31 (Estimated)

PRIMARY OUTCOMES:
functional capacity | 6 months
  functional capacity change measured with 6-minute walk test

SECONDARY OUTCOMES:
functional capacity | 12 months
  functional capacity change measured with 6-minute walk test
NT-proBNP | 6 months
  N-terminal pro-B-type natriuretic peptide levels
hsCRP | 6 months
  high-sensitivity C-reactive protein
pulmonary congestion | 6 and 12 months
  assessed by ultrasound detection of B-lines
physical activity | 6 and 12 months
  average daily step count measured over 7 days by ActiGraph
depression | 6 and 12 months
  assessed with the Beck Depression Inventory-II
health-related quality of life | 6 and 12 months
  assessed with the 36-Item Short Form Health Survey (SF-36)
self-efficacy | 6 and 12 months
  assessed with the Czech version of the General Self-Efficacy scale (DOVE)
body mass index | 6 and 12 months
  calculated by dividing the body weight (kg) by the square of the height (m2)
waist circumference | 6 and 12 months
  recorded with a measurement tape to the nearest 0.1 cm
hip circumference | 6 and 12 months
  recorded with a measurement tape to the nearest 0.1 cm
Meta-Analysis Global Group in Chronic Heart Failure (MAGGIC) Risk Score | 6 and 12 months
  method to predict survival in heart failure patients

CONTACTS AND LOCATIONS:
Overall Officials: Jan Belohlavek, Ass. Prof., Principal Investigator — Charles University, Czech Republic
Locations (1):
- General University Hospital in Prague, Prague, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vetrovsky T, Siranec M, Parenica J, Griva M, Stastny J, Precek J, Pelouch R, Bunc V, Linhart A, Belohlavek J. Effect of a 6-month pedometer-based walking intervention on functional capacity in patients with chronic heart failure with reduced (HFrEF) and with preserved (HFpEF) ejection fraction: study protocol for two multicenter randomized controlled trials. J Transl Med. 2017 Jul 3;15(1):153. doi: 10.1186/s12967-017-1257-x. PMID 28673328